CLINICAL TRIAL: NCT01022073
Title: CSP #468F - Long Term Study of Deep Brain Stimulation for Parkinson's Disease: A Longitudinal Follow-Up Study of the VA/NINDS CSP #468 Cohort
Brief Title: Follow Up Study for Treatment of Parkinson's Disease With Deep Brain Stimulation
Acronym: CSP#468F
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 468F
Record Dates: First submitted 2009-11-25; First posted 2009-12-01 (Estimated); Results first posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-05

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation; Subthalamic Nucleus; Globus Pallidus; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Globus Pallidus interna Group: Cohort of subjects who received DBS-GPi as part of the CSP 468 intervention trial, and still have their device working and in place.
- Subthalamic Nucleus Group: Cohort of subjects who received DBS-STN as part of the CSP 468 intervention trial, and still have their device working and in place.

SUMMARY:
Follow up of patients enrolled in CSP 468, a study of deep brain stimulation treatment for Parkinson's disease

DETAILED DESCRIPTION:
Parkinson's disease (PD), the second most prevalent neurodegenerative disease (after Alzheimer's disease), affects more than a million Americans and is a common condition in the Veteran population. Although there is currently no cure for the disease, many of the symptoms of the disease can be effectively managed with medications and with deep brain stimulation (DBS). This study seeks to build upon the original CSP#468 protocol by providing an efficient long-term follow-up study. The objectives of this study are to:

determine whether the motor benefits of deep brain stimulation persist beyond two years of follow-up in patients with Parkinson's disease; determine whether the target of stimulation (GPi vs. STN) affects the durability of long-term motor improvement; define the impact of DBS on long-term function and quality of life in patients with Parkinson's disease; identify clinical features that predict favorable or unfavorable long-term outcome; and describe the long-term performance of the DBS devices, including device durability, device explanation rate, neurostimulator replacement frequency, and changes in stimulation parameters to achieve optimum symptom control.

ELIGIBILITY:
Inclusion Criteria:

* Participant in CSP#468
* Available and willing to be followed-up according to study protocol

Exclusion Criteria:

* DBS device explanted or permanently turned off without anticipated resumption of DBS therapy.

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's Disease who were enrolled in CSP 468, and received DBS.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2010-06; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J. Marks, MD, Study Chair — San Francisco VA Medical Center, San Francisco, CA
Locations (12):
- United States (12):
  - UCLA-University of California at Los Angeles(904), Los Angeles, California
  - San Francisco-University of California at San Francisco(905), San Francisco, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California
  - VA Medical Center, Portland, Portland, Oregon
  - Portland-Oregon Health & science University(906), Portland, Oregon
  - VA Medical Center, Philadelphia, Philadelphia, Pennsylvania
  - Philadelphia-University of Pennsylvania Health System(901), Philadelphia, Pennsylvania
  - Houston-Methodist Hospital(903), Houston, Texas
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Richmond-Medical college of Virginia(902), Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
We can share the data based on the VA approved Data Use Agreement(DUA)

REFERENCES:
- [Derived] Ostrem JL, Luo P, Weaver FM, Follett K, Rothlind J, Galifianakis NB, Lai EC, Bronstein J, Duda J, Holloway K, Sarwar A, Brodsky M, Chung K, Spindler M, Reda D, Snodgrass A, Moy C, Huang G, Wei Y, Marks WJ Jr; CSP 468F Study Group. 10-year clinical outcomes of subthalamic nucleus versus pallidal deep brain stimulation for Parkinson's disease: VA/NINDS CSP #468F. Front Neurol. 2026 Jan 16;16:1728999. doi: 10.3389/fneur.2025.1728999. eCollection 2025. PMID 41626017

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The original study CSP #468 visits were completed in October 2008, and the kick-off meeting for the follow-up study was held on April 26-28, 2010. Out of the total randomized 299 participants in the main study of CSP#468, 156 participants enrolled in this follow-up study. Subject recruitment started in August 2010 and ended in September 2011.
Pre-assignment Details: This is follow-up study from the original study CSP#468.
Period: Overall Study
Arm/Group | Globus Pallidus Interna Group | Subthalamic Nucleus Group
Started | 86 | 70
Completed | 67 | 52
Not Completed | 19 | 18

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Globus Pallidus Interna Group | Subthalamic Nucleus Group | Total
Number analyzed (Participants) | 86 | 70 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (8.4) | 58.6 (7.9) | 59.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 75 | 58 | 133
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 84 | 66 | 150
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 86 | 70 | 156
Married Status [Number; unit: participants]
  Married | 65 | 49 | 114
  Single/Never Married | 4 | 2 | 6
  Seperated | 1 | 0 | 1
  Divorced | 16 | 19 | 35
Living with Family [Number; unit: participants]
  Alone | 6 | 9 | 15
  With Family | 75 | 57 | 132
  With Non-Family | 5 | 3 | 8
  Nursing | 0 | 1 | 1
Family history of Parkinson's Disease [Number; unit: participants]
  yes | 19 | 20 | 39
  no | 67 | 50 | 117
Years since Parkinson's Disease diagnosis [Mean (Standard Deviation); unit: years] | 11.4 (4.7) | 11.4 (5.2) | 11.4 (4.9)
Years on Parkinson's Disease medications [Mean (Standard Deviation); unit: years] | 11.0 (4.7) | 10.6 (4.7) | 10.8 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Off-medication/On-stimulation Motor Function Score of the Unified Parkinson's Disease Rating Scale (UPDRS Part III)
Description: The primary outcome measure for the comparison of GPi deep brain stimulation (DBS) to STN DBS is the motor function score of the Unified Parkinson's Disease Rating Scale (UPDRS Part III) measured while the patient is off medications and on stimulation at follow-up visits post surgery. UPDRS Part III has 14 items assessing motor skills including facial expression and speech, tremors, rigidity, posture, gait, and bradykinesia. Left and right sides (arms, legs, and hands) are assessed separately for seven of the functions. A summary score ranging from 0 to 108 is generated by adding the 14 specific motor function responses. The motor function (UPDRS part III) assessments are done by turning on the stimulation with and without taking PD medications (on/off) at each in-person visit. The higher the value, the worse the outcome.
Time Frame: The change score of UPDRS Part III from baseline to 9 years post surgery
Population: Patients had completed the 9 year follow-up post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Globus Pallidus Interna Group | Subthalamic Nucleus Group
Number analyzed (Participants) | 50 | 28
units on a scale | -8.2 (14.6) | -9.1 (14.2)
Statistical Analysis 1: Comparison: Globus Pallidus Interna Group vs Subthalamic Nucleus Group; Test type: Superiority or Other; p = 0.808, t-test, 2 sided; This analysis is based on the completers. We are working on the imputation methods to account for the missing data and will revise results later

ADVERSE EVENTS:
Description: This study only collected study related serious adverse events given that there is no intervention.
Arm/Group | Globus Pallidus Interna Group | Subthalamic Nucleus Group
Serious Adverse Events (participants affected / at risk) | 2/86 | 2/70
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Globus Pallidus Interna Group (N=86) | Subthalamic Nucleus Group (N=70)
Elective Hospitalization (Surgical and medical procedures) | 2 (2) | 2 (2) — Elective hospitalization are not medical events and are only scheduled to facilitate a safe study visit for the participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes